CLINICAL TRIAL: NCT01683097
Title: Assessing Patient Understanding and Factors That Govern Advanced Directives and End of Life Discussion
Brief Title: Patient Understanding of End of Life Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Partners in Internal Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SVH 1195
Record Dates: First submitted 2012-07-25; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Advance Directives; Resuscitation Orders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Questionnaire
- Intervention (Experimental): Standardized explanation followed by questionnaire
  Interventions: Other: Standardized explanation

INTERVENTIONS:
Other: Standardized explanation — Standardized explanation provided on code status, advance directives and end of life care
  Arms: Intervention

SUMMARY:
This study aims at assessing factors that affect patient choices for end of life care. 300 patients would be assigned either to a control arm (questionnaire alone) or intervention arm (standardized explanation+ questionnaire). Our intervention is a standardized explanation which explains what code status, advance directive and end of life care mean. Based on patient responses, factors that affect choices of code status would be analyzed. We will also evaluate if a standardized explanation improves patient understanding of end of life issues. This would be determined by generating a composite score of correct responses to a subset of objective questions in the questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Admitted to regular nursing floor

Exclusion Criteria:

* altered mental status
* admitted in ICU
* positive screening for depression
* terminal illness defined as life expectancy< 100 days
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Composite score of correct responses | Patients interviewed within 48 hours of admission, questionnaire adminsitered at the time of interview
  Patients in both arms were administered a questionnaire, that assessed demographics, subjective questions as well as a set of objective questions designed to assess patient understanding of code status. The responses to the objective questions were scored and the composite score of correct responses was used as a marker of patient understanding. Patients in the control arm were administered the questionnaire alone. Patients in the intervention arm first received our standard explanation, and were then administered the questionnaire

SECONDARY OUTCOMES:
Compare differences in demographic, medical, social and associated factors on patient choice of code status | Patients interviewed within 48 hours of admission, questionnaire adminsitered at the time of interview

CONTACTS AND LOCATIONS:
Overall Officials: George Abraham, MD, Principal Investigator — Saint Vincent Hospital; Kriti Mittal, MD, Principal Investigator — Saint Vincent Hospital
Locations (1):
- Saint Vincent Hospital, Worcester, Massachusetts, United States